CLINICAL TRIAL: NCT03146273
Title: A Pharmacokinetic Crossover Comparison Study of Absorption Characteristics of Two Multivitamin Mineral Formulations (Gel vs. Tablet/Capsule)
Brief Title: Study of Absorption Characteristics of Two Multivitamin Mineral Formulations (Gel vs. Tablet/Capsule)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galilee CBR (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: SSPA-17-1
Record Dates: First submitted 2017-05-06; First posted 2017-05-09 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Vitamin Deficiency
MeSH Terms: conditions — Avitaminosis | interventions — Geritol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet (Active Comparator): The tablet/capsule will be administered as a single dose of Multivitamins in tablet after 12 hours of fasting. The participants will be monitored during 6 hours for the level of minerals and Multivitamin minerals in the blood, adverse events and vital signs. The results will be used for the AUC calculation of the absorption in order to compare with the Gel administration absorption.
  Interventions: Dietary Supplement: Multivitamins
- Gel (Active Comparator): The gel will be administrated to the same group of patients in the single dose of Multivitamins in gel after 12 hours of fasting. The participants will be monitored during 6 hours for the level of minerals and Multivitamin minerals in the blood, adverse events and vital signs. The results will be used for the AUC calculation of the absorption in order to compare with the Tablet administration absorption.
  Interventions: Dietary Supplement: Multivitamins

INTERVENTIONS:
Dietary Supplement: Multivitamins — After the study product administration blood tests will be performed in order to calculate the AUC for each mineral and vitamin - Vit A Vit E Folic Acid Vit C Calcium Magnesium
  After the washout period, the same procedure will be done for the additional formulation of the multivitamins.

SUMMARY:
This clinical study is designed to evaluate difference in the AUC of the absorption of Multivitamin and minerals defined in the protocol

DETAILED DESCRIPTION:
This clinical study is designed to evaluate difference in the AUC of the absorption of Multivitamin and minerals:

1. Tablet/capsule administration - up to 20 healthy volunteers will be recruited to the study. The tablet/capsule will be administered as a single dose after 12 hours of fasting. The participants will be monitored during 6 hours for the level of minerals and Multivitamin minerals in the blood, adverse events and vital signs.
2. Gel administration - the gel will be administrated to the same group of patients in the single dose after 12 hours of fasting. The participants will be monitored during 6 hours for the level of minerals and Multivitamin minerals in the blood, adverse events and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female and aged 18-65 years
* BMI - 19-24
* Subject is not pregnant and is not nursing
* Signed Informed Consent Form

Exclusion Criteria:

* Current use of multivitamin or mineral complexes (washout of 4 days before Visit 2 is permitted)
* Participants with known vitamins or mineral deficiencies
* Diabetes Type II
* Smoking
* Subjects who have undergone surgery within the last 3 months.
* Subjects with a clinically significant (during last 3 months) infectious, immune-mediated or active malignant disease.
* Subjects who are receiving an elemental diet or parenteral nutrition.
* Subjects who are treated with insulin.
* Women with childbearing potential unless surgically sterile or using adequate contraception (either IUD, oral or Depo-provera contraceptive, or barrier plus spermicide); pregnant or breastfeeding mothers.
* Subjects who will be unavailable for the duration of the trial, who are unlikely to be compliant with the protocol, or who are felt to be unsuitable by the Investigator for any other reason.
* Known sensitivity to any ingredients in the study product
* History of addiction or drug abuse
* Alcoholic regular use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2017-06-10 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Mean fractional absorption | 6 hours
  A comparison of mean fractional absorption of the two Multivitamin mineral formulations (gel vs. tablet/capsule).

SECONDARY OUTCOMES:
Absorption rate | 6 hours
  A comparison of absorption rate across the two Multivitamin mineral formulations (gel vs. tablet/capsule).

CONTACTS AND LOCATIONS:
Locations (1):
- Israel, Tel Aviv, Central District, Israel

IPD SHARING:
Plan to Share IPD: No
The study results will be published.